CLINICAL TRIAL: NCT02439450
Title: A Phase 1b/2 Study of Viagenpumatucel-L (HS-110) in Combination With Multiple Treatment Regimens in Patients With Non-Small Cell Lung Cancer (The "DURGA" Trial)
Brief Title: A Study of Combination Therapies With Viagenpumatucel-L (HS-110) in Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Heat Biologics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS110-102
Record Dates: First submitted 2015-05-04; First posted 2015-05-08 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-10

CONDITIONS: Non-small Cell Lung Cancer
Keywords: lung; cancer; gp96; vaccine; immunotherapy; Heat Biologics; Nivolumab; checkpoint inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Nivolumab; pembrolizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 5: Viagenpumatucel-L + Nivolumab CPI Naive (Experimental): Patients naïve to checkpoint inhibitor (CPI) therapy will receive a combination of weekly HS-110 administered as 5 intradermal 0.1 mL injections at a dose of 1 × 107 viable cells/ 0.5 mL for 18 weeks and bi-weekly nivolumab infusions. After 18 weeks of treatment, patients will continue on monotherapy standard of care nivolumab until confirmed disease progression or unacceptable toxicity, whichever occurs first. After the completion of 18 weeks of combination therapy, patients may receive either nivolumab dosing schedule listed in the current approved package insert (every 2 weeks or every 4 weeks) per Investigator discretion.
  Interventions: Biological: Viagenpumatucel-L; Drug: Nivolumab
- Arm 6: Viagenpumatucel-L + pembrolizumab (Experimental): HS-110 dosing to be initiated at/before the start of the 3rd maintenance treatment cycle, or within 19 weeks of front-line pembrolizumab monotherapy. Patients will receive a combination of weekly HS-110 administered as 5 intradermal 0.1 mL injections at a dose of 1 × 107 viable cells/0.5 mL for 13 weeks in combination with SOC pembrolizumab every 3 weeks. Following the 13-week priming period, HS-110 injections will be administered for boosting every 3 weeks in combination with SOC pembrolizumab until confirmed disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Biological: Viagenpumatucel-L; Drug: Pembrolizumab
- Arm 5: Viagenpumatucel-L + Nivolumab CPI Progressor (Experimental): Patients with prior checkpoint inhibitor (CPI) therapy will receive a combination of weekly HS-110 administered as 5 intradermal 0.1 mL injections at a dose of 1 × 107 viable cells/ 0.5 mL for 18 weeks and bi-weekly nivolumab infusions. After 18 weeks of treatment, patients will continue on monotherapy standard of care nivolumab until confirmed disease progression or unacceptable toxicity, whichever occurs first. After the completion of 18 weeks of combination therapy, patients may receive either nivolumab dosing schedule listed in the current approved package insert (every 2 weeks or every 4 weeks) per Investigator discretion.
  Interventions: Biological: Viagenpumatucel-L; Drug: Nivolumab
- Arm 6: Viagenpumatucel-L + pembrolizumab + pemetrexed (Experimental): HS-110 dosing to be initiated at/before the start of the 3rd maintenance treatment cycle, or within 19 weeks of front-line pembrolizumab monotherapy. Patients will receive a combination of weekly HS-110 administered as 5 intradermal 0.1 mL injections at a dose of 1 × 107 viable cells/0.5 mL for 13 weeks in combination with SOC pembrolizumab + pemetrexed every 3 weeks. Following the 13-week priming period, HS-110 injections will be administered for boosting every 3 weeks in combination with SOC pembrolizumab + pemetrexed until confirmed disease progression or unacceptable toxicity, whichever occurs first.
  Interventions: Biological: Viagenpumatucel-L; Drug: Pembrolizumab; Drug: Pemetrexed

INTERVENTIONS:
Biological: Viagenpumatucel-L — Vaccine derived from irradiated human lung cancer cells genetically engineered to continually secrete gp96-Ig
  Other Names: HS-110
Drug: Nivolumab — Nivolumab 240mg IV q2weeks for 18 weeks or until disease progression or unacceptable toxicity. After the completion of 18 weeks of combination therapy, patients may receive either nivolumab dosing schedule listed in the current approved package insert (every 2 weeks or every 4 weeks) per Investigator discretion.
  Other Names: Opdivo
  Arms: Arm 5: Viagenpumatucel-L + Nivolumab CPI Naive; Arm 5: Viagenpumatucel-L + Nivolumab CPI Progressor
Drug: Pembrolizumab — The recommended dose of KEYTRUDA (pembrolizumab) is 200 mg administered as an intravenous infusion over 30 minutes every 3 weeks until disease progression, unacceptable toxicity, or up to 24 months in patients without disease progression.
  Other Names: Keytruda
  Arms: Arm 6: Viagenpumatucel-L + pembrolizumab; Arm 6: Viagenpumatucel-L + pembrolizumab + pemetrexed
Drug: Pemetrexed — The recommended dose of ALIMTA (pemetrexed) when administered with carboplatin and pembrolizumab for the initial treatment of NSCLC in patients with a creatinine clearance (calculated by Cockcroft-Gault equation) of 45 mL/min or greater is 500 mg/m2 administered as an intravenous infusion over 10 minutes prior to carboplatin on Day 1 of each 21-day cycle for 4 cycles. Pembrolizumab should be administered prior to ALIMTA when given on the same day.
  Other Names: Alimta
  Arms: Arm 6: Viagenpumatucel-L + pembrolizumab + pemetrexed

SUMMARY:
This study will test whether vaccination with viagenpumatucel-L combined with strategies to modulate the immune response is safe for patients with non-small cell lung adenocarcinoma or squamous cell carcinoma for incurable or metastatic disease.

DETAILED DESCRIPTION:
This study will test whether vaccination with viagenpumatucel-L combined with strategies to modulate the immune response is safe for patients with non-small cell lung adenocarcinoma or squamous cell carcinoma for incurable or metastatic disease. These methods collectively use the body's immune system to target the patient's own tumor. Immunosuppression hinders that response, and may develop in NSCLC patients in a variety of ways, such as activation of checkpoint pathways in the tumor microenvironment. Drugs that disrupt checkpoint molecule signaling like anti-PD-1 monoclonal antibodies nivolumab, may release this brake on the immune system. Tumor expression of PD-L1 plays an important role in patient response to checkpoint inhibitors; in general, clinical response to checkpoint inhibitors requires tumor expression of PD-L1 and presence of Tumor Infiltrating Lymphocytes (TIL). Combining viagenpumatucel-L with anti-PD-1 agents may enhance the vaccine's anti-tumor activity while prolonging or increasing the efficacy of the checkpoint inhibitor.

ELIGIBILITY:
INCLUSION CRITERIA:

* Non-small cell lung adenocarcinoma or squamous cell carcimona
* At least one site of measurable disease by RECIST 1.1
* Arm 5: Received at least one prior line of therapy, but no more than three prior lines of therapy, for incurable (i.e. unresectable) or metastatic NSCLC. Up to one prior line of FDA-approved checkpoint inhibitor therapy is permitted (must have received at least 4 months of treatment) --OR--
* Arm 6: Received front line immunotherapy (with or without chemotherapy) for incurable or metastatic NSCLC and did not progress clinically or radiographically per RECIST 1.1 at the most recent imaging assessment, and will begin maintenance immunotherapy with standard of care pembrolizumab ± pemetrexed.
* Life expectancy ≥18 weeks
* Arm 5: Disease progression at study entry --OR--
* Arm 6: Documented Stable Disease, Partial Response, Complete Response (SD/PR/CR) per RECIST 1.1 after a minimum of 9 to 12 weeks of front line immunotherapy (with or without chemotherapy).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Central nervous system (CNS) metastases may be permitted but must be treated and neurologically stable
* Adequate laboratory parameters
* Willing and able to comply with the protocol and sign informed consent
* Female patients who are of childbearing potential and fertile male patients must agree to use an effective form of contraception throughout study participation
* Willing to provide archival or fresh tumor biopsy at Screening, and fresh tumor biopsy at Week 10 when feasible.
* Arm 5: Suitable for treatment with nivolumab per package insert --OR--
* Arm 6: Suitable for front line maintenance treatment with pembrolizumab ± pemetrexed per the current approved package inserts.

EXCLUSION CRITERIA:

* Arm 5: Received systemic anticancer therapy within 21 days prior to first dose of study drug
* Human immunodeficiency virus (HIV), hepatitis B or C, or severe/uncontrolled infections or concurrent illness, unrelated to the tumor, requiring active therapy
* Any condition requiring concurrent systemic immunosuppressive therapy
* Known immunodeficiency disorders, either primary or acquired
* Known leptomeningeal disease
* Active malignancies within 12 months with the exception of those with a negligible risk of metastasis or death treated with expected curative outcome
* Pregnant or breastfeeding
* Prior participation in a clinical study of viagenpumatucel-L (HS-110)
* Administration of a live vaccine within 30 days prior to first dose of study drug
* Active, known or suspected autoimmune disease
* Significant cardiovascular disease
* Refractory to prior immunotherapy (clinical or radiographic progression after 12 weeks or less of immunotherapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Morgensztern, MD, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (16):
- United States (16):
  - University of Arizona Cancer Center, Tucson, Arizona
  - UC San Diego, La Jolla, California
  - BRRH Lynn Cancer Institute, Boca Raton, Florida
  - Memorial Cancer Institute, Pembroke Pines, Florida
  - Horizon Oncology Research, Lafayette, Indiana
  - Ashland-Bellefonte Cancer Center, Ashland, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Washington University School of Medicine, St Louis, Missouri
  - New York Oncology Hematology, Albany, New York
  - Winthrop Hospital, Mineola, New York
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Virginia Cancer Specialists, Fairfax, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 5: Viagenpumatucel-L + Nivolumab CPI Naïve: Patients naïve to CPI therapy will receive a combination of weekly HS-110 administered as 5 intradermal 0.1 mL injections at a dose of 1 × 107 viable cells/ 0.5 mL for 18 weeks and bi-weekly nivolumab infusions. After 18 weeks of treatment, patients will continue on monotherapy standard of care nivolumab until confirmed disease progression or unacceptable toxicity, whichever occurs first. After the completion of 18 weeks of combination therapy, patients may receive either nivolumab dosing schedule listed in the current approved package insert (every 2 weeks or every 4 weeks) per Investigator discretion.
  Viagenpumatucel-L: Vaccine derived from irradiated human lung cancer cells genetically engineered to continually secrete gp96-Ig
  Nivolumab: Nivolumab 240mg IV q2weeks for 18 weeks or until disease progression or unacceptable toxicity. After the completion of 18 weeks of combination therapy, patients may receive either nivolumab dosing schedule listed in the current approved package insert (every 2 weeks or every 4 weeks) per Investigator discretion.
- Arm 5: Viagenpumatucel-L + Nivolumab CPI Progressor: Patients with prior CPI therapy will receive a combination of weekly HS-110 administered as 5 intradermal 0.1 mL injections at a dose of 1 × 107 viable cells/ 0.5 mL for 18 weeks and bi-weekly nivolumab infusions. After 18 weeks of treatment, patients will continue on monotherapy standard of care nivolumab until confirmed disease progression or unacceptable toxicity, whichever occurs first. After the completion of 18 weeks of combination therapy, patients may receive either nivolumab dosing schedule listed in the current approved package insert (every 2 weeks or every 4 weeks) per Investigator discretion.
  Viagenpumatucel-L: Vaccine derived from irradiated human lung cancer cells genetically engineered to continually secrete gp96-Ig
  Nivolumab: Nivolumab 240mg IV q2weeks for 18 weeks or until disease progression or unacceptable toxicity. After the completion of 18 weeks of combination therapy, patients may receive either nivolumab dosing schedule listed in the current approved package insert (every 2 weeks or every 4 weeks) per Investigator discretion.
Period: Overall Study
Arm/Group | Arm 5: Viagenpumatucel-L + Nivolumab CPI Naïve | Arm 5: Viagenpumatucel-L + Nivolumab CPI Progressor | Arm 6: Viagenpumatucel-L + Pembrolizumab | Arm 6: Viagenpumatucel-L + Pembrolizumab + Pemetrexed
Started | 47 | 68 | 2 | 4
Completed | 21 | 24 | 0 | 0
Not Completed | 26 | 44 | 2 | 4
Not completed — Adverse Event | 4 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Death | 3 | 0 | 0 | 1
Not completed — Progressive Disease | 18 | 41 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Arm 6: Viagenpumatucel-L + Pembrolizumab +/- Pemetrexed: HS-110 dosing to be initiated at/before the start of the 3rd maintenance treatment cycle, or within 19 weeks of front-line pembrolizumab monotherapy. Patients will receive a combination of weekly HS-110 administered as 5 intradermal 0.1 mL injections at a dose of 1 × 107 viable cells/0.5 mL for 13 weeks in combination with SOC pembrolizumab ± pemetrexed every 3 weeks. Following the 13-week priming period, HS-110 injections will be administered for boosting every 3 weeks in combination with SOC pembrolizumab ± pemetrexed until confirmed disease progression or unacceptable toxicity, whichever occurs first.
  Viagenpumatucel-L: Vaccine derived from irradiated human lung cancer cells genetically engineered to continually secrete gp96-Ig
  Pembrolizumab: The recommended dose of KEYTRUDA (pembrolizumab) is 200 mg administered as an intravenous infusion over 30 minutes every 3 weeks until disease progression, unacceptable toxicity, or up to 24 months in patients without disease progression.
  Pemetrexed: The recommended dose of ALIMTA (pemetrexed) when administered with carboplatin and pembrolizumab for the initial treatment of NSCLC in patients with a creatinine clearance (calculated by Cockcroft-Gault equation) of 45 mL/min or greater is 500 mg/m2 administered as an intravenous infusion over 10 minutes prior to carboplatin on Day 1 of each 21-day cycle for 4 cycles. Pembrolizumab should be administered prior to ALIMTA when given on the same day.
- Total: Total of all reporting groups
Arm/Group | Arm 5: Viagenpumatucel-L + Nivolumab CPI Naïve | Arm 5: Viagenpumatucel-L + Nivolumab CPI Progressor | Arm 6: Viagenpumatucel-L + Pembrolizumab | Arm 6: Viagenpumatucel-L + Pembrolizumab +/- Pemetrexed | Total
Number analyzed (Participants) | 47 | 68 | 2 | 4 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8.9) | 67 (9.1) | 70 (12.7) | 70 (5.1) | 67 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 37 | 1 | 3 | 67
  Male | 21 | 31 | 1 | 1 | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 11 | 0 | 0 | 15
  White | 42 | 54 | 2 | 4 | 102
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Frequency of Treatment Emergent Adverse Events (TEAEs) as Assessed by CTCAE v4.03.
Description: The number and percent of patients with a given TEAE will be summarized overall and by system organ class and preferred term by treatment group. The number and percent of patients with TEAEs will be tabulated by maximum severity.
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5: Viagenpumatucel-L + Nivolumab CPI Naive | Arm 6: Viagenpumatucel-L + Pembrolizumab | Arm 5: Viagenpumatucel-L + Nivolumab CPI Progressor | Arm 6: Viagenpumatucel-L + Pembrolizumab + Pemetrexed
Number analyzed (Participants) | 47 | 68 | 2 | 4
Participants | 47 | 66 | 2 | 4

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Arm 5: Viagenpumatucel-L + Nivolumab CPI Naïve | Arm 5: Viagenpumatucel-L + Nivolumab CPI Progressor | Arm 6: Viagenpumatucel-L + Pembrolizumab | Arm 6: Viagenpumatucel-L + Pembrolizumab + Pemetrexed
All-Cause Mortality (participants affected / at risk) | 39/47 | 60/68 | 2/2 | 3/4
Serious Adverse Events (participants affected / at risk) | 13/47 | 16/68 | 0/2 | 1/4
Other Adverse Events (participants affected / at risk) | 47/47 | 66/68 | 2/2 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 5: Viagenpumatucel-L + Nivolumab CPI Naïve (N=47) | Arm 5: Viagenpumatucel-L + Nivolumab CPI Progressor (N=68) | Arm 6: Viagenpumatucel-L + Pembrolizumab (N=2) | Arm 6: Viagenpumatucel-L + Pembrolizumab + Pemetrexed (N=4)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 5: Viagenpumatucel-L + Nivolumab CPI Naïve (N=47) | Arm 5: Viagenpumatucel-L + Nivolumab CPI Progressor (N=68) | Arm 6: Viagenpumatucel-L + Pembrolizumab (N=2) | Arm 6: Viagenpumatucel-L + Pembrolizumab + Pemetrexed (N=4)
Anaemia (Blood and lymphatic system disorders) | 7 (10) | 7 (11) | 0 (0) | 2 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 8 (8) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7) | 10 (10) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 11 (11) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 11 (11) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 6 (6) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 13 (13) | 23 (26) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 4 (6) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 4 (4) | 6 (6) | 0 (0) | 2 (2)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3) | 7 (7) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 4 (5) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 4 (4) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 7 (11) | 7 (9) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (5) | 7 (10) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 4 (4) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 4 (4) | 10 (10) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 3 (4) | 2 (2) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 11 (11) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (9) | 7 (7) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 4 (4) | 9 (9) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 8 (8) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 8 (10) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (5) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 6 (8) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 6 (6) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 9 (11) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 6 (6) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 6 (6) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 10 (11) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 12 (14) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 8 (9) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 5 (5) | 0 (0) | 0 (0)
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (7) | 11 (11) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5) | 0 (0) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 4 (6) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 7 (7) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 6 (8) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT02439450/Prot_SAP_000.pdf